CLINICAL TRIAL: NCT03200834
Title: Comparison of D2 vs D3 Lymph Node Dissection for Right Colon Cancer (RICON)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: G.V. Bondar Republican Cancer Center (Other)
Collaborators: Donetsk National Medical University (Other); I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2017-03-25; First posted 2017-06-27 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Colon Cancer
Keywords: Right colon cancer; D3 dissection; complete mesocolic excision; Hemicolectomy
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D2 lymph node dissection for right colon cancer (Active Comparator): Hemicolectomy for right colon cancer with D2 lymph node dissection
  Interventions: Procedure: Right Hemicolectomy with D2 lymph node dissection
- D3 lymph node dissection for right colon cancer (Experimental): Hemicolectomy for right colon cancer with D3 lymph node dissection
  Interventions: Procedure: Right Hemicolectomy with D3 lymph node dissection

INTERVENTIONS:
Procedure: Right Hemicolectomy with D2 lymph node dissection — Remove right part of colon with lymph node dissection №201, №202, №211, №212 (if present), №221,№222 (Japanese classification).
  Arms: D2 lymph node dissection for right colon cancer
Procedure: Right Hemicolectomy with D3 lymph node dissection — Remove right part of colon with lymph node dissection №201, №202, № 203, №211, №212 (if present), №213 (if present) №221,№222, №223 (for hepatic flexure and proximal part of transverse colon cancer)(Japanese classification).
  Arms: D3 lymph node dissection for right colon cancer

SUMMARY:
Comparing different method of surgical technique D2 lymph node dissection vs D3 for right colon cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Agreement of the patient to participate in trial
2. Colon cancer (only adenocarcinoma )
3. The tumor located between the cecum and the right 1/3 of transverse colon
4. Tumors T3,Т4а,b N0-2 (II-III stages)
5. Tolerance of chemotherapy
6. ECOG 0-2

Exclusion Criteria:

1. Patients with distant metastases
2. Tumors T1-2 (I stage)
3. Complications of tumor (perforation and full bowel obstruction)
4. Previous radiotherapy or chemotherapy
5. Synchronous or metachronous tumors
6. Women during Pregnancy or breast feeding period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2029-01-03 (Estimated); Study Completion 2029-01-03 (Estimated)

PRIMARY OUTCOMES:
5-year survival | Up to 5 years post-operative
  death from any cause

SECONDARY OUTCOMES:
morbidity | within the first 30 days after surgery
  postoperative complications
mortality | within the first 30 days after surgery
  death after surgery
Disease free survival 5 years after initial surgery | Up to 5 years post-operative
  local and distant metastasis during 5 years after operation

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Balaban, PhD, Study Director — M.Gorky Donetsk National Medical University
Locations (1):
- G.V. Bondar Republican Cancer Center, Donetsk, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Balaban V, Mutyk M, Bondarenko N, Zolotukhin S, Sovpel O, Sovpel I, Zykov D, Rublevskiy I, Klochkov M, Prado AP, He M, Tsarkov P. Comparison of D2 vs D3 lymph node dissection for RIght COloN cancer (RICON): study protocol for an international multicenter open-label randomized controlled trial. Trials. 2024 Jul 2;25(1):438. doi: 10.1186/s13063-024-08269-5. PMID 38956698